CLINICAL TRIAL: NCT01709097
Title: Compliance/Adherence After Kidney Transplant, With or With Out an Electronic Drug Dispenser(Med-O-Wheel™), Karolinska University Hospital.
Brief Title: Compliance/Adherence After Kidney Transplant, With or With Out Med-O-Wheel™.
Acronym: C/A
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: Addoz (Other); Roche Pharma AG (Industry); Tele2Sverige AB (Unknown)
Responsible Party: Principal Investigator, Gunnar Tydén, Professor, Karolinska University Hospital
Other Study IDs: Dnr 2011/471-31/4
Record Dates: First submitted 2012-10-16; First posted 2012-10-17 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-08

CONDITIONS: Medication Adherence; Compliance; Medication Nonadherence; Communication; Transplant; Failure, Kidney
Keywords: Adherence; Compliance; Kidney Transplant Recipient; An electronic drug dispenser; The Portal
MeSH Terms: conditions — Medication Adherence; Patient Compliance; Communication

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- With Med-O-Wheel™: Kidney Transplant Recipient with Med-O-Wheel™
- With out Med-O-Wheel™: Kidney Transplant Recipient with out Med-O-Wheel™

SUMMARY:
Background:

Adherence to the immunosuppressive drug regimen is critical to the outcome after an organ transplant. Patients need to take their prescribed medications and attend their appointments with the doctor.

Based on previous studies in other European countries, the cost of non-compliance after organ transplantation in Sweden is >SEK 35 million/year.

Patients who lose their graft both lose quality of life and have decreased expected survival; moreover, retransplantation may be hampered by new HLA antibodies.

Question:

The primary question is whether Med-O-Wheel™ can improve compliance to the prescribed medication regimen in renal transplant patients.

Methods and materials:

All kidney transplant patients at Karolinska University Hospital, Huddinge, will be given information about the study and will then be asked to participate. Participants will be randomized into two arms, one arm with and one with out Med-O-Wheel™. The 80 included patients will be closely monitored for 1 year regarding intake of prescribed medications.

Med-O-Wheel™ is an electronic medication dispenser that records the date and time of each occasion when the patient takes medications from the dispenser. It has a SIM card and text messaging capabilities.

Addoz Portal™ is a web-based application that makes it possible to monitor and analyse medication intake. Each event in the medication dispenser is registered in the portal, which communicates with the care provider/support person by text message, e-mail or telephone.

Significance of the study:

In the future it may be possible to improve compliance in transplant patients. In particular, patients will feel secure since they will receive confirmation through the portal that they are taking their medications safely and accurately.

DETAILED DESCRIPTION:
Study objectives:

To investigate whether Med-O-Wheel™ can improve -

1. adherence to medication regimens,
2. adherence to appointments at the outpatient clinic, and
3. treatment outcome in renal transplant patients. Methodology

Study design:

Open, prospective, descriptive, randomized study.

Primary research question:

Can Med-O-Wheel™ improve adherence to the prescribed medication regimen in renal transplant patients?

Efficacy parameters:

P-Creatinine, concentrations of medication (B-tacrolimus, B-cyclosporine, B-sirolimus, P/S-mycophenolate, B-TPMT-metabolites) and age(years).

Addoz Portal for Med-O-Wheel™. Study-specific questionnaire to survey patient discomfort relating to compliance and adherence.

Safety parameters:

Med-O-Wheel™ and Addoz Portal™ is a CE-approved product with a guarantee for continuous operation. Karolinska University Laboratory is an accredited testing laboratory.

Volunteer population

Subjects:

All patients about to undergo renal transplantation at Karolinska University Hospital.

Number: 80 patients (40 patients with Med-O-Wheel™, 40 patients with out Med-O-Wheel™).

Time frame First patient included: Juni 2011. Last patient included: Juli 2012. Last patient completed: Juli 2013.

ELIGIBILITY:
Subject is eligible for the study if the following apply:

* Receiving a kidney transplant from a deceased or living donor in Karolinska University Hospital
* Capable of understanding the purpose of the study, fully informed and having written informed consent (signed Informed Consent has been obtained)

No study-specific exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Kidney Transplant Recipients in Karolinska University Hospital
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2011-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Can Med-O-Wheel™ improve adherence to the prescribed medication regimen in renal transplant patients? | 2013

CONTACTS AND LOCATIONS:
Overall Officials: Jarmo Henriksson, SC, RN, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829